CLINICAL TRIAL: NCT03259698
Title: Optimizing the Delivery of HIV Post-exposure Prophylaxis: A Randomized Controlled Trial of Text Messaging Support and Physician to Nurse Task-shifting
Brief Title: Optimizing the Delivery of HIV nPEP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTN 287
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM 1 = TEXT MESSAGING SUPPORT (Experimental): PEP will be delivered by ID physician and participants will receive weekly text message "check-ins" and optional automated text appointment reminders via the WelTel system.
  Interventions: Drug: nPEP; Behavioral: Text Messaging Support
- ARM 2 = NO TEXT MESSAGING SUPPORT (Experimental): PEP will be delivered according to the standard of care by an infectious diseases physician. Participants will not receive text message reminders or "check-in".
  Interventions: Drug: nPEP
- ARM 3 = NURSE-LED nPEP (Experimental): PEP will be delivered by a sexual health clinic nurse operating under a medical directive.
  Interventions: Drug: nPEP; Other: Nurse-Led nPEP
- ARM 4 = ID PHYSICIAN-LED nPEP, (Active Comparator): PEP will be delivered according to the standard of care by an infectious diseases physician.
  Interventions: Drug: nPEP

INTERVENTIONS:
Drug: nPEP — Participants will receive Bictegravir/emtricitabine/tenofovir alafenamide 50/200/25mg (Biktarvy®) one tablet once daily as study drug to complete a 28 day course of PEP.
  Other Names: Biktarvy; Bictegravir/emtricitabine/tenofovir alafenamide; BIC/FTC/TAF
Behavioral: Text Messaging Support — Text messaging support service ('WelTel'): community-based counselors will provides standardized weekly 'check-in' messages during the participants 12-week course of nPEP follow-up. Participants in the text-message arm will also have the option of receiving generic non-specific automated text reminders of their upcoming appointments in the form of "Don't forget about tomorrow".
  Arms: ARM 1 = TEXT MESSAGING SUPPORT
Other: Nurse-Led nPEP — nPEP follow-up is provided by nurse-led care at a local sexual health clinic instead of a hospital-based ID physician.
  Arms: ARM 3 = NURSE-LED nPEP

SUMMARY:
Despite decades of traditional prevention efforts based on behavior change and condom use, Ontario has seen over 700 new HIV infections annually over the past 10 years. Post-exposure prophylaxis (PEP) is one such approach, in which uninfected persons use 28 days of antiretroviral medications (ARVs) shortly after an HIV exposure to minimize the risk of acquiring HIV. PEP is highly efficacious, is considered a standard of care intervention based on medical and ethical grounds, and is supported by treatment guidelines. Yet several implementation challenges have limited its clinical and public health impact in Ontario, where no formal PEP policy exists. Our proposal seeks to optimize two aspects of delivering PEP for sexual exposures (nPEP). Results will inform the development of a standardized approach to nPEP both province-wide and elsewhere.

Thus study has pragmatic, multicenter randomized controlled trial using a 2x2 factorial design to determine whether the proportion of nPEP patients that successfully complete follow-up:

1. is higher among those receiving mobile phone-based text messaging support than among those receiving standard care; and
2. is non-inferior among those receiving care from a sexual health clinic nurse compared to those receiving hospital-based physician care.

The prospective, randomized, non-blinded, 2x2 factorial trial that will enroll 318 study participants in Toronto. In Intervention A, we will randomize half of study participants to a text messaging support service ('WelTel'), in which a trained, community-based counselor provides standardized weekly 'check-in' messages during their 12-week course of PEP follow-up. The other half will receive standard care, which does not include any form of active outreach or reminders outside of scheduled appointments. In Intervention B, we will randomize half of participants to receive nurse-led care for PEP follow-up at a local sexual health clinic; the other half will receive standard care by a hospital-based ID physician. The specific activities for each follow-up visit will be clearly defined in a medical directive. In keeping with Ontario legislation on medical directives, nurses will review cases with their authorizing physician or nurse practitioner on a routine basis.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older
2. Be known or presumed to be HIV-uninfected at baseline
3. Be initiated on PEP by a healthcare provider in the past six days for a sexual exposure to a known or suspected HIV-infected source
4. STAGE 1 only: Own a mobile phone with text messaging capabilities on which they are willing to potentially receive messages from the text messaging service
5. Be capable of communicating verbally and via text in English
6. Be planning to continue their follow-up locally or be willing to have follow-up study visits conducted remotely; either by telephone or via an encrypted video conferencing system (such as Zoom for healthcare).
7. Be referred to a sexual assault center and provided with necessary counselling and support services if presented for nPEP following sexual assault.

Exclusion Criteria:

1. Creatinine clearance <30 mL/min (using Cockcroft-Gault formula)
2. Enrolled in any other clinical trial of an HIV prevention intervention
3. Prior participation in this clinical trial for a previous episode of nPEP
4. Known co-infection with chronic hepatitis B at enrollment
5. Current or planned pregnancy or breastfeeding
6. Use of a medication whose co-administration with Biktarvy is contraindicated (dofetilide, carbamazepine, oxcarbazepine, phenobarbital, phenytoin, rifampin, rifampicin, rifabutin, rifapentine, modafinil, dexamethasone, metformin, St. John's Wort)
7. Concomitant use of HIV pre-exposure prophylaxis (PrEP)
8. Stage 2 only: Concomitant use of any non-prescription medication, supplement, vitamin or natural remedy which the patient is unwilling to discontinue during Biktarvy® administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Self-reported completion of a full course of PEP medications and receipt of a final HIV test result from their nPEP provider 12 weeks after the index exposure | 12 weeks
  Determined by patient completion of acceptability questionnaire and evidence of HIV test result

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability of TAF/FTC/ELV/cobi-based nPEP] | 12 weeks
  Collection of adverse events
Completion of each scheduled follow-up activity (blood tests and clinic visits) | 12 weeks
  Measured by study visit attendance on CRFs
Diagnosis of incident HIV | 12 weeks
  Determined through laboratory analysis of blood, urine and mucosal swab samples
Sexually transmitted infections (gonorrhea, chlamydia, syphilis, hepatitis B and C) | 12 weeks
  Determined through laboratory analysis of blood sample
Self-reported sexual risk-taking behaviour | 12 weeks
  The following activities will be captured in a questionnaire: number of unprotected vaginal/anal sex acts, and for men who have sex with men, score on a HIV risk index (based on the validated HIRI-MSM)
Numbers and types of linkages made by PEP providers to other forms of healthcare | Week 12
  1. Number of participants referred to psychiatry/mental health services and
  2. Number of participants referred to addictions/substance services
Patient satisfaction with their PEP experience | 12 weeks
  Collected using a patient survey
Inquiries from participants to the PEP provider outside of scheduled follow-up | 12 weeks
  the number of times participants contacted their healthcare provider outside of scheduled follow-up
PEP-related referrals for physician consultation | 12 weeks
  Number of times a participant randomized to the nurse-led arm had to be referred to a physician; captured on the sexual health clinic documentation.

OTHER OUTCOMES:
Assessment of cost on heathcare system | Week 12
  Prospective collection of cost data during the trial to inform a future health economic analysis from the perspective of the healthcare system.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell HS Tan, MD, FRCPC, PhD, Principal Investigator — Unity Health Toronto; Isaac I Bogoch, MD, FRCPC, MSc, Principal Investigator — Toronto General Hospital
Locations (3):
- Canada (3):
  - HIV Prevention Clinic (Toronto General Hospital), Toronto, Ontario
  - Positive Care Clinic (St. Michael's Hospital), Toronto, Ontario
  - Crossways Sexual Health Clinic (TPH), Toronto

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730